CLINICAL TRIAL: NCT00264199
Title: The Effect of 48 Hours GLP-1 Infusion on Left Ventricular Function, Exercise Capacity, Insulin Sensitivity and Substrate Metabolism in Patients With Chronic Heart Failure
Brief Title: Effect of 48 Hours of Treatment With the Natural Peptide-Hormone GLP-1 in Patients With Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: University of Aarhus (Other); Aarhus University Hospital (Other)
Responsible Party: Mads Halbirk, Aarhus University Hospital, Skejby
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20050048
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Heart Failure, Congestive
Keywords: Chronic Congestive heart failure; Ischemic heart disease; insulin resistance
MeSH Terms: conditions — Heart Failure; Myocardial Ischemia; Insulin Resistance | interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: GLP-1
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: GLP-1 — iv. by weight (1.0 pmol/kg/min )
  Arms: 1
Drug: placebo — same rate of infusion as GLP-1
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether 48 hours of glucagon-like-peptide-1 (GLP-1) infusion can improve heart function and alter substrate metabolism in non-diabetic patients with heart failure.

DETAILED DESCRIPTION:
Heart failure is a major complication in patients with ischemic heart disease. It has been shown that many of these patients have areas of viable myocardium that are not effectively contributing to heart function.

Further, chronic congestive heart failure is associated with some degree of insulin resistance in both skeletal and cardiac muscle.

GLP-1 is a naturally occurring peptide hormone that acts as an incretin and has been intensively studied by many groups in association with type II diabetes and it has clearly shown its glucose lowering potential with very little risk of hypoglycemia in several trials.

Recently GLP-1 has been shown to improve cardiac function in dogs with pace-induced cardiomyopathy, and in an open-labeled study it did improve cardiac function in patients with acute myocardial infarctions.

Comparison: 48 hours of treatment with intravenous GLP-1 compared to placebo. Effect on global and regional left ventricular function, exercise capacity, insulin sensitivity and substrate metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Chronic congestive heart failure
* Ischemic heart disease

Exclusion Criteria:

* Diabetes
* Exercise limiting disease other than heart failure
* Congenital heart disease
* Arterio-venous shunts
* Renal failure
* Valvular heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-12; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Effect on global left ventricular function | at baseline and after 48 hours of intervention
Effect on regional left ventricular function | at baseline and after 48 hours of intervention
Effect on exercise capacity | at baseline and after 48 hours of intervention
Effect on 6 minute walk test | at baseline and after 48 hours of intervention
Effect on insulin sensitivity | after 48 hours of intervention
Effect on substrate metabolism at whole-body level and in the fore-arm | after 48 hours of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hans Erik Bøtker, MD, Principal Investigator — Afdeling B, Skejby Hospital
Locations (1):
- Afdeling B, Skejby Hospital, Aarhus, Denmark